CLINICAL TRIAL: NCT02678143
Title: A Pilot Study of Nonmyeloablative Conditioning for Mismatched Hematopoietic Stem Cell Transplantation for Severe Sickle Cell Disease
Brief Title: Nonmyeloablative Conditioning for Mismatched Hematopoietic Stem Cell Transplantation for Severe Sickle Cell Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Closed early due to competing studies
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201602019
Record Dates: First submitted 2016-02-04; First posted 2016-02-09 (Estimated); Last update posted 2022-02-14 (Actual); Status verified 2022-01

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Alemtuzumab; Cyclophosphamide; Mycophenolic Acid; Sirolimus; fludarabine; fludarabine phosphate; Whole-Body Irradiation; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Recipients (Experimental): * The recipient of one antigen mismatch unrelated HSCT will begin the preparative regimen on Day -7. Alemtuzumab on Days -7, -6, -5, -4, and -3, cyclophosphamide on Days -4 and -3, and 300 cGy of total body irradiation (TBI) on Day -2.
  * The recipient of haplo-SCT will begin the preparative regimen on Day -7. Alemtuzumab on Days -7, -6, -5, -4, and -3, fludarabine on Days -7, -6, -5, -4, and -3, cyclophosphamide on Days -4 and -3, and 400 cGy of TBI on Day -2.
  * For both types of HSCT, the frozen peripheral blood stem cells will be thawed and infused on Day 0 per institutional guidelines. GVHD prophylaxis will consist of cyclophosphamide on Days +3 and + 4, mycophenolate mofetil (MMF) three times a day on Days +5 through +35 then tapered off over 1 week provided there is no evidence of GVHD, and sirolimus starting on Day +5 and continuing for one year. Sirolimus can be tapered at one year only if donor T-cell chimerism reaches more than 50% in the absence of GVHD.
  Interventions: Drug: Alemtuzumab; Drug: Cyclophosphamide; Drug: Mycophenolate mofetil; Drug: Sirolimus; Drug: Fludarabine; Radiation: Total body irradiation; Procedure: Hematopoietic stem cell transplant

INTERVENTIONS:
Drug: Alemtuzumab
  Other Names: Campath
Drug: Cyclophosphamide
  Other Names: Revimmune; Clafen; Cytoxan; Neosar
Drug: Mycophenolate mofetil
  Other Names: CellCept
Drug: Sirolimus
  Other Names: Rapamune
Drug: Fludarabine
  Other Names: Oforta; Fludara
Radiation: Total body irradiation
  Other Names: TBI
Procedure: Hematopoietic stem cell transplant

SUMMARY:
The aim of this study is to evaluate the overall safety and feasibility of using haploidentical or one antigen mismatch unrelated hematopoietic stem cell transplant (HSCT) for adult patients with severe sickle cell disease (SCD) who undergo a non-myeloablative preparative regimen consisting of total body irradiation (TBI), cyclophosphamide and alemtuzumab (and fludarabine for haplo-SCT only) and graft vs. host disease (GvHD) prophylaxis consisting of post-transplant cyclophosphamide (PT-Cy), mycophenolate mofetil (MMF), and sirolimus. The investigators anticipate that this approach will expand the donor pool and offer a safe and less toxic curative intervention.

ELIGIBILITY:
Recipient Inclusion Criteria:

* Age greater than or equal to 19 years.
* Diagnosis of sickle cell disease (HB SS, SC, or SBeta-thal(0)); confirmed by hemoglobin electrophoresis, high-performance liquid chromatography, DNA testing when necessary or both.
* At high risk for disease-related morbidity or mortality, defined by having at least one of the following manifestations (A-E):

  * A: Clinically significant neurologic event (stroke) or any neurological deficit lasting > 24 hours.
  * B: History of two or more episodes of acute chest syndrome (ACS) in the 2-year period preceding enrollment despite the institution of supportive care measures including hydroxyurea.
  * C: Three or more pain crises per year in the 2-year period preceding referral (required intravenous pain management in the outpatient or inpatient hospital setting) despite the institution of supportive care measures including hydroxyurea.
  * D: Administration of regular RBC transfusion therapy, defined as receiving 8 or more transfusions per year for ≥ 1 year to prevent vaso-occlusive clinical complications (i.e. pain, stroke, acute chest syndrome, and priapism).
  * E: Pulmonary hypertension (defined as tricuspid regurgitant jet velocity (TRV) ≥2.5 m/s at baseline (without vaso-occlusive crisis)
* Any one of the below complications not ameliorated by hydroxyurea at the maximum tolerated dose for at least 6 months:

  * Vaso-occlusive crises with more than 1 hospital admission per year while on maximal tolerated dose of hydroxyurea
  * Acute chest syndrome occurring while on hydrox*Eyurea
  * Age greater than or equal to 19 years.
* Availability of one antigen mismatched unrelated or haploidentical related donor
* Cerebral MRI/MRA within 30 days prior to initiation of transplant conditioning. If there is clinical or radiologic evidence of a recent neurologic event (such as stroke or transient ischemic attack) subjects will be deferred for at least 6 months with repeat cerebral MRI/MRA to ensure stabilization of the neurologic event prior to proceeding to transplantation.
* Ability to comprehend and willing to sign an informed consent

Recipient Exclusion Criteria:

* Detectable antibody to ABO, Rh, or other red blood cell antigen of their donors
* Presence of donor specific antibodies detected by donor specific antibody screen (if using product from a haploidentical donor).
* Karnofsky/Lansky performance score < 60
* Evidence of uncontrolled bacterial, viral, or fungal infections (currently taking medication and progression of clinical symptoms) within one month prior to starting the conditioning regimen. Patients with fever or suspected minor infection should await resolution of symptoms before starting the conditioning regimen.
* Poor cardiac function defined as left ventricular ejection fraction < 40%.
* Poor pulmonary function defined as FEV1 and FVC < 40% predicted or diffusing capacity of the lung for carbon monoxide (DLCO) < 40% (corrected for hemoglobin)
* Poor liver function defined as direct bilirubin > 2x upper limit of normal for age and alanine aminotransferase (ALT) and aspartate aminotransferase (AST) > 5 times upper limit of normal.
* Poor kidney function defined by creatinine clearance < 70mL/min.
* HIV-positive.
* Unwillingness to use approved contraception method from time of biologic assignment until discontinuation of all immunosuppressive medications.
* Demonstrated lack of compliance with prior medical care (determined by referring physician).
* Pregnant or breastfeeding.
* Diagnosis of any debilitating medical or psychiatric illness that would preclude giving informed consent or receiving optimal treatment and follow-up.

Donor Selection:

* Must be one antigen mismatched unrelated donor or first-degree relative who shares at least one HLA haplotype with the recipient.
* Must not have SCD or another hemoglobinopathy.
* In good health based on institutional standards.
* Weight ≥ 20kg.
* If donor is < 18 years old must have ability to give informed assent based on institutional standards for pediatric donors.
* Able to undergo peripheral blood stem cell mobilization with G-CSF
* Hemoglobin S ≤ 50%.
* HIV-1&2 antibody, HTLV-I&II antibody, HBV and HCV sero-negative.

  * Note: When more than one donor is available, the donor with the lowest number of HLA allele mismatches will be chosen, unless there is HLA cross-match incompatibility or a medical reason to select otherwise, in which case donor selection is the responsibility of the PI, in consultation with the immunogenetics laboratory. In cases where there is more than one donor with the least degree of mismatch, donors will be selected based on the most favorable combination of (i) HLA compatibility in cross-match testing, (ii) ABO compatibility, (iii) CMV status and (iv) non-inherited maternal antigens (NIMAs) mismatching.
  * HLA crossmatching (in order of priority)

    * Mutually compatible (no cross-matching antibodies)
    * Recipient non-cross-reactive with donor, donor cross-reactive with recipient
    * Mutually cross-reactive
  * ABO compatibility (in order of priority)

    * Compatible
    * Major incompatibility
    * Minor incompatibility
    * Major and minor incompatibility
  * CMV negative donor is preferred
  * NIMA mismatched donor is preferred

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-04-26 (Actual); Primary Completion 2020-04-03 (Actual); Study Completion 2021-11-16 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of treatment regimen as measured by grade 3, 4, and 5 toxicities | From time of consent through Day 180 (estimated to be 6 months)
  -The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for all toxicity reporting.

SECONDARY OUTCOMES:
Feasibility of treatment regimen as measured by accrual | Completion of study accrual (up to 10 years)
Feasibility of treatment regimen as measured by patient compliance to treatment and follow-up | Up to 2 years
  -Patient compliance to treatment and follow-up will be measured by how many appointments the patient misses
Rate of engraftment | Day 100
Incidence of acute graft-versus-host disease | Up to Day 140
  -Acute GVHD grade will be accessed using MAGIC criteria
Incidence of transplant related mortality | Up to 2 years
  -Death that results from a transplant procedure-related complication (e.g. infection, organ failure, hemorrhage, GVHD), rather than from relapse of the underlying disease or an unrelated cause.
Incidence of engraftment failure | Day 100
  -Engraftment failure (GF) will be determined as the proportion of patients having undetectable DNA of donor origin on at least 2 occasions no less than 1 week apart at day +100.
Overall survival rate | 1 year
  -Overall survival (OS) is defined as the date from transplant to death or last follow-up.
Overall survival rate | 2 years
  -Overall survival (OS) is defined as the date from transplant to death or last follow-up.
Event-free survival rate | 1 year
  -Event-free survival (EFS) is defined as the date of transplant to the date of an event or last follow-up. An event is defined as toxicity (graft failure, death) or a disease-related event (stroke, acute chest syndrome, pain crisis) with full recipient-type hemoglobin on hemoglobin electrophoresis for patients with sickle cell disease.
Event-free survival rate | 2 years
  -Event-free survival (EFS) is defined as the date of transplant to the date of an event or last follow-up. An event is defined as toxicity (graft failure, death) or a disease-related event (stroke, acute chest syndrome, pain crisis) with full recipient-type hemoglobin on hemoglobin electrophoresis for patients with sickle cell disease.

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Schroeder, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu